CLINICAL TRIAL: NCT00477945
Title: A Phase I Trial of Clofarabine in Combination With High-Dose Etoposide and Cyclophosphamide and Autologous Peripheral Blood Stem Cell Transplantation for Patients With High-Risk or Refractory Non-Hodgkin's Lymphoma
Brief Title: Phase I Trial of Clofarabine in Combo w/ HD Etoposide & Cyclophosphamide and APBSCT for Pts w/ High-Risk or Refractory NHL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Collaborators: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Indiana University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0704-29 IUCRO-0187
Record Dates: First submitted 2007-05-22; First posted 2007-05-24 (Estimated); Last update posted 2014-09-11 (Estimated); Status verified 2014-09

CONDITIONS: Non Hodgkin's Lymphoma
Keywords: Non Hodgkin's Lymphoma; High Risk or Refractory Non Hodgkin's Lymphoma; APBSCT; clofarabine
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Clofarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: clofarabine — Cohort N Clofarabine (mg/m2/day)
  1. 3-6 30
  2. 3-6 40
  3. 3-6 50
  4. 3-6 60
  5. 6-10 70

SUMMARY:
This is a phase I trial to determine the maximum tolerated dose (MTD) of clofarabine in a combination with high-dose etoposide and cyclophosphamide. This is an initial step in developing a novel myeloablative preparative regimen for autologous hematopoietic stem cell transplantation (ASCT). While this phase I trial will initially develop the regimen in patients with refractory disease, it is expected that it will find its best application in patients with less advanced disease.

DETAILED DESCRIPTION:
All patients will receive the same doses of etoposide and cyclophosphamide. The dose of clofarabine will be escalated in successive cohorts of patients. Using a standard dose escalation design, successive cohorts of 3 patients will be treated with escalating doses of clofarabine (see Section 5.5 below). At the MTD (or highest dose-level if the MTD is not reached), the cohort will be expanded to 10 patients to better investigate correlative studies and give some preliminary idea of efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Documentation of disease. Patients must have one of the following disease types:

   * Diffuse large cell non-Hodgkin's lymphoma, mediastinal B-cell lymphoma, or peripheral T-cell lymphoma that is:

     * Primary refractory (achievement less than complete response)
     * Relapsed and refractory (achievement less than a partial response) to at least a single salvage therapy
   * Relapsed or primary refractory Follicular lymphoma (FL) with a high FL International Prognostic Index.
   * Large cell transformation of lymphoma from a more indolent lymphoma (e.g., follicular, marginal zone, etc.)
   * Mantle cell lymphoma that is:

     * Primary Refractory (achievement less than complete response)
     * Relapsed (regardless of chemosensitivity of relapsed disease)
2. Patients who received prior autologous stem cell transplantation are not eligible.
3. Patient age 18-70 years
4. Performance status ECOG 0-1
5. Required baseline laboratory values:

   * LVEF > 45% corrected
   * DLCO > 50% of predicted value (corrected for hemoglobin)
   * Serum creatinine ≤ 2.0 mg/dl or estimated creatinine clearance of ≥60 ml/min
   * Bilirubin < 1 x upper limit of normal value.
   * AST and ALT < 1 x upper limit of normal value.
6. Signed written informed consent. Patient must be capable of understanding the investigational nature of the investigational nature, potential risks and benefits of the study, and able to provide valid informed consent

Exclusion Criteria:

1. No active infection. Patients with active infections requiring oral or intravenous antibiotics are not eligible for enrollment until resolution of infection.
2. No HIV disease. Patients with immune dysfunction are at a significantly higher risk of infection from intensive immunosuppressive therapies.
3. Non-pregnant and non-nursing. Treatment under this protocol would expose a fetus to significant risks. Women of childbearing potential should have a negative pregnancy test prior to study entry. Women and men of reproductive potential should agree to use an appropriate method of birth control throughout their participation in this study due to the teratogenic potential of the therapy utilized in this trial. Appropriate methods of birth control include oral contraceptives, implantable hormonal contraceptives (Norplant®), or double barrier method (diaphragm plus condom).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-05; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose (MTD) of clofarabine in association with high-dose etoposide and cyclophosphamide followed by ASCT in patients with refractory lymphoma malignancies. | 1 yr

SECONDARY OUTCOMES:
Assessment of the toxicity of the combination of clofarabine, and high-dose etoposide and cyclophosphamide-- Describe engraftment kinetics-- Describe the response rate-- Describe relapse rate and event-free survival-- Assess clofarabine p | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sherif Farag, MD, PhD, Principal Investigator — Indiana University
Locations (1):
- Indiana University Cancer Center, Indianapolis, Indiana, United States